CLINICAL TRIAL: NCT04974385
Title: Comparison of Liposomal Bupivacaine Versus Non-liposomal Bupivacaine for Total Shoulder Arthroplasty: a Prospective, Double-blinded, Noninferiority Trial
Brief Title: Liposomal Bupivacaine Versus Non-liposomal Bupivacaine for Total Shoulder Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, D. Aric Elmer, MD, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSR210190
Record Dates: First submitted 2021-07-03; First posted 2021-07-23 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal Bupivacaine (Experimental): Experimental group will receive ISNB with admixed LB (10 mL) and 0.5% bupivacaine (10 mL) total of 20 mL.
  Interventions: Drug: Liposomal bupivacaine; Drug: Bupivacaine
- Non-liposomal Bupivacaine (Active Comparator): Comparator group will receive ISNB with 20 mL of 0.5% non-liposomal bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Validate the analgesic efficacy of admixed LB + bupivacaine compared with plain bupivacaine when injected for ISNB for total shoulder arthroplasty.
  Other Names: Exparel
  Arms: Liposomal Bupivacaine
Drug: Bupivacaine — Active comparator as standard of care.

SUMMARY:
The objective of this study is to validate the analgesic efficacy of admixed Liposomal bupivacaine (LB) + bupivacaine compared with plain bupivacaine when injected for interscalene nerve block (ISNB) for total shoulder arthroplasty (TSA). We hypothesize that admixed LB will be non-inferior to plain bupivacaine in terms of postoperative opioid consumption following TSA. The primary outcome of this study will be opioid consumption over the first 72 hours following surgery. Secondary outcomes will include: pain scores, opioid-related adverse events, block related adverse events, pain related phone calls, pain related ED visits and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Undergoing total shoulder arthroplasty
* Willing and able to sign consent form to participate in study

Exclusion Criteria:

* < 18 years of age
* Unwilling or unable to sign consent form to participate in study
* Allergy to local anesthetic
* Medical contraindication to interscalene nerve block
* Chronic opioid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | 72 hours postoperative
  Morphine equivalents used during first 72 hours after surgery

SECONDARY OUTCOMES:
Numeric Rating Scale Reported Pain Scores | 72 hours postoperative
  Patient reported pain scores using the numeric rating scale from 0 to 10 where 0 means no pain and 10 means worst possible pain
Nerve Block Related Adverse Events | 72 hours postoperative
  Any adverse event determined to be caused as a result of having a nerve block to include but not limited to toxicity, allergic reaction, nerve injury.
Patients with Additional, Unanticipated Pain Related Medical Encounters | 72 hours postoperative
  Any unanticipated, unplanned, pain related phone calls to surgeon or anesthesiologist for rescue pain treatment, pain related emergency department visits or primary care physician visits for pain treatment
Patient Reported Satisfaction with Postoperative Pain Control Using the Numeric Rating Scale | 72 hours postoperative
  Patient reported satisfaction with their postoperative pain control using the numeric rating scale from 0 to 10 where 0 means completely dissatisfied and 10 means completely satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Donald A Elmer, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Medical Center, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No